CLINICAL TRIAL: NCT00154544
Title: Identification of Biomarkers Associated With Human Hepatocellular Carcinoma by PROTEOMEX
Brief Title: Searching for the Liver Cancer-Related Biomarkers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9261701419; NSC 93-2314-B-002-228
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2005-12-20 (Estimated); Status verified 2003-12

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Hepatocellular carcinoma (HCC) has been the leading cause of cancer death in Taiwan. About 6000-8000 people died of this cancer every year in Taiwan. Though regular sonographic examination can early detect small HCC and there are many therapeutic modalities for HCC, the therapeutic results remains unsatisfactory. Though Alpha-fetoprotein (AFP) and des-γ-carboxy prothrombin (DCP) are used as the tumor markers for diagnosis of HCCs, these two markers are not good enough for the early detection of small HCCs. To improve the survival, further investigations of the early diagnostic markers are still needed. In this current project, we applied the proteomic method to identify the HCC biomarkers.

DETAILED DESCRIPTION:
Cell lines Hep3B and Huh7 HCC cell lines will be cultured in (Dulbecco's modified Eagle medium) DMEM containing 10% fetal calf serum and incubated at 37 C in 5% CO2 incubator. The rationale of using HCC cell line instead of clinical HCC samples is that HCC tissues are heterogeneous and might contain some non-HCC cells. The cell will be harvested when cells reach 95% confluence.

Sera collection 20 mL of venous 20 mL of venous blood was collected from 20 HBV-related HCC and 20 HCV-related HCC patients before treatment. The venous blood was allowed to clot, centrifuged at 800 g for 5 min, and serum was aliquoted and stored at -80 0C. Control sera were obtained from 20 HBV carriers without HCC, 20 chronic hepatitis C patients without HCC, and 10 normal subjects without liver diseases.

Two-dimensional gel electrophoresis using patients' sera for immunoblotting will be done. Spots of interest will be identified by delayed extraction matrix-assisted laser desorption ionization.

ELIGIBILITY:
Inclusion Criteria:

* hepatocellular carcinoma

Exclusion Criteria:

* multiple cancers

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2004-08

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Hung Chen, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan